CLINICAL TRIAL: NCT05208567
Title: London Valvular Heart Disease and Reduced Ejection Fraction Detection in a Multi-ethnic Community Using Cardiac Ultrasound
Acronym: LOVE
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 292737
Record Dates: First submitted 2022-01-21; First posted 2022-01-26 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Heart Valve Diseases; Left Ventricular Dysfunction
MeSH Terms: conditions — Heart Valve Diseases; Ventricular Dysfunction, Left | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Cardiac Ultrasound Scan - using an abbreviated protocol

SUMMARY:
Heart Valve Disease and Heart failure contribute to 25% of hospital emergency admissions while heart failure alone has become one of the most common causes for hospitalisation in people over the age of 65. The burden of disease is likely to be high in a multi-ethnic community but there is a paucity of data. Management of heart valve disease requires appropriate surveillance and timely surgery. Similarly heart failure management requires treatment with medications aimed at slowing prevention of symptoms and preventing premature death. The NHS long term plan priorities early detection and treatment of valve disease and heart failure in order to reduce the burden on emergency services and improve the health of the population.

Diagnosis is made using cardiac ultrasound, however staff with the required skills-set are critically limited in the community.

The investigators will train non-expert staff within primary care to perform abbreviated cardiac ultrasound to detect heart valve disease or heart failure. This will be opportunistic scanning to reduce healthcare footfall.

All scans will be reviewed by an expert and the investigators will use the anonymised data to develop machine learning tools to begin working with academic partners to develop tools that can improve the reliability of diagnosis from ultrasound.

The investigators hope to identify the proportion with the above conditions in a multi-ethnic community and assess the feasibility of developing a program where staff can be trained for community detection, streamlined referrals can be created bridging the gap between primary and secondary care, reducing hospital emergency admissions, while ensuring patients are managed optimally.

ELIGIBILITY:
Inclusion Criteria:

- Greater or equal to 65 years old

Exclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease or Vascular Dementia
* Palliative Care patients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who are ≥65yrs old who are attending their GP practice for an appointment will be studied. All patients with pre-existing diagnoses of valvular heart disease or Left Ventricular Dysfunction will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-08-02 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants within a North East London community over the age of 65yrs old with Valvular Heart Disease, as assessed by Cardiac Ultrasound | 12 months
  Participants will be recruited while attending their routine health check at their GP practice and consented for a cardiac ultrasound to identify Valvular Heart Disease
Number of participants within a North East London community over the age of 65yrs old with Left Ventricular Systolic Dysfunction as assessed by Cardiac Ultrasound | 12 months
  Participants will be recruited while attending their routine health check at their GP practice and consented for a cardiac ultrasound to identify Left Ventricular Systolic Dysfunction.
Diagnostic accuracy in identifying heart valve disease or left ventricular systolic dysfunction using abbreviated echocardiography following training protocols. | 12 months
  Trainees will be taught how to perform and interpret focussed cardiac ultrasound scans, their interpretations and performance will be measured against an expert's and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomews Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided